CLINICAL TRIAL: NCT02049502
Title: The Use of Fecal Microbiota Transplantation in Patients With Ulcerative Colitis-associated Pouchitis
Brief Title: FMT in Ulcerative Colitis-Associated Pouchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia O. Shaffer (Other)
Responsible Party: Sponsor-Investigator, Virginia O. Shaffer, M.D., Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071015
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Ulcerative Colitis Associated Pouchitis
Keywords: ulcerative colitis; fecal microbiota transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fecal microbiota transplant (Experimental): fecal microbiota transplant
  Interventions: Biological: biologically active human fecal microbiota; Procedure: sigmoidoscopy

INTERVENTIONS:
Biological: biologically active human fecal microbiota — instillation of biologically active human fecal microbiota material via flexible sigmoidoscopy
Procedure: sigmoidoscopy

SUMMARY:
The purpose of this study is to test whether Fecal Microbiota Transplant (FMT) is a safe and effective treatment for people who have Ulcerative Colitis and have had an ileal pouch anastomosis.

Ulcerative colitis (UC) is a type of inflammatory bowel disease (IBD) that may be caused by a person's immune system responding in an unusual way to bacteria normally found in the gut. Studies have shown that the gut bacteria in people with ulcerative colitis (UC) are different from the gut bacteria in people without ulcerative colitis (UC). Often, people with ulcerative colitis (UC) have fewer types of bacteria in their gut which can change the way that person's immune system works.

This study is for people who have had a proctocolectomy with an ileal pouch anastomosis (IPAA) to treat ulcerative colitis (UC). More than 50% of people who have had an IPAA will develop a condition called pouchitis. Pouchitis is short or long-term inflammation of the ileal pouch that was created in order to store waste from your intestines. Patients with pouchitis are being asked to take part in this study.

Currently, antibiotics, probiotics and prebiotics are used to treat pouchitis. However, it has been shown that probiotics are not very helpful once the patient stops taking them. In addition, antibiotics may cause unfavorable side effects. Fecal microbiota transplantation (FMT) is being studied as another form of treatment for patients with active pouchitis. Fecal microbiota transplantation (FMT) or "stool transplant" involves receiving a single fecal enema from someone who has volunteered to donate their stool.

There are two purposes of this research study:

1. To see whether or not fecal microbiota transplantation (FMT) is a useful treatment for patients with ulcerative colitis (UC) associated pouchitis
2. To study the changes within the bacteria in the gut in patients with pouchitis (before and after study treatment) using stool, blood and urine samples

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 18 to 65 years
* ulcerative colitis-associated pouchitis
* patients of Emory Clinic and/or Emory University Hospital

Exclusion Criteria:

* Age <18 years or >65 years of age
* Exposure to immunosuppressive therapy (defined as steroid, etanercept, or anti-tumor necrosis factor (TNF)agents) within 1 month prior to enrollment
* Concomitant Clostridium difficile infection
* Suspected Crohn's disease
* Documented active infection of any kind
* Patients on anti-coagulant therapy, with platelet count less than 50,000, significant anemia with hemoglobin less than 7 or those with other conditions that place them at increased risk of bleeding
* Absolute neutrophil count (ANC) less than 1000 or history of opportunistic infection
* Administration of investigational drug within one month prior to planned FMT
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia O. Shaffer, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiota Transplant: fecal microbiota transplant
  biologically active human fecal microbiota: instillation of biologically active human fecal microbiota material via flexible sigmoidoscopy
  sigmoidoscopy
Period: Overall Study
Arm/Group | Fecal Microbiota Transplant
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Improvement of Pouchitis Symptoms
Description: Improvement of clinical pouchitis symptoms based on the clinical component of the modified pouchitis disease activity index (mPDAI) without relapse. These components include: stool frequency (number of stools), rectal bleeding, fecal urgency or abdominal cramps, or fever (temperature >37.8C).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 8
Participants | 2

2. Secondary Outcome: Number of Patients With Favorable Microbiota Profile
Description: 16s ribosomal gene sequencing and metabolomic profile of the gut microbiota
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Fecal Microbiota Transplant
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (N=8)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Increase in stool frequency (Gastrointestinal disorders) | 1 (1)
Fever (Reproductive system and breast disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT02049502/Prot_SAP_000.pdf